CLINICAL TRIAL: NCT03513497
Title: IFI16 is a Periodontitis Modulating Protein
Acronym: IFI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18-0291; 1K01DE027087-01 (NIH)
Record Dates: First submitted 2018-04-19; First posted 2018-05-01 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-05

CONDITIONS: Severe Periodontitis; Acute Inflammatory Response
Keywords: Teeth; Periodontal disease; acute inflammatory response; stent-induced biofilm overgrowth; periodontal pathogens
MeSH Terms: conditions — Periodontitis; Periodontal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periodontal Profile Class (PPC-A) (Experimental): Periodontally healthy participants (PPC-A) and participants with mild disease (PPC-B) will wear customized acrylic mouthguard only during tooth brushing for 21 days.
  Interventions: Other: Customized acrylic mouthguard
- Periodontal Profile Class (PPC-G) (Experimental): Participants with severe periodontal disease (PPC-G) and participants with posterior disease (PPC-E) will wear customized acrylic mouthguard only during tooth brushing for 21 days.
  Interventions: Other: Customized acrylic mouthguard

INTERVENTIONS:
Other: Customized acrylic mouthguard — Customized acrylic mouthguards extended to cover approximately 2 mm over gingival margins will be fabricated for each subject. Stents will form a seal and rest on the gingiva, but will be relieved on the tooth and tissue side except for the occlusal surfaces to avoid disturbing plaque or gingival tissues. Acrylic stents will cover the area in one sextant where no brushing and flossing teeth is to occur for 21 days.
  Other Names: intraoral stent

SUMMARY:
To characterize the expression of Interferon gamma inducible protein 16 (IFI16) and Absent in melanoma 2 (AIM2) in gingival tissues in an inflammatory response using an acrylic mouthguard (also referred to as a stent) induced bacteria overgrowth method.

Participants: A maximum of 72 Adult subjects will be recruited from the patients, students and staff at the University of North Carolina, as well as the general population in or near Chapel Hill NC.

Procedures (methods):

Medical history, demographics, (height/weight), urine based pregnancy test, vital signs (to include blood pressures, and pulse) standard dental clinical measures (to include plaque index, gingival index, bleeding on probing, and clinical attachment level), alginate impressions taken for fabrication of an acrylic stent (mouthguard), 2 gingival biopsies, 2 subgingival (below the gumline) plaque samples, and Scaling Root planing (SRP)/or adult prophylaxis

DETAILED DESCRIPTION:
A total of 72 subjects will be enrolled. Specifically, a sufficient number of adults 18 years and older will be screened until 36 healthy (PPC-A) subjects and 36 subjects with severe periodontal disease (PPC-G) will be enrolled. Eligibility for study participation will be determined during the screening session. Barring dropout, subject participation will include 1 to 8 visits lasting over a maximum period of 42 days. The last 3 visits (visit 5-8) will depend on the individual need of the subject for providing SRP. Clinical data and medical history data will be collected at the screening visit to ascertain eligibility. All subjects will have dental plaque and a gingival biopsy collected at baseline. Enrolled subjects will be included in an experimental gingivitis model Stent-Induced Biofilm Overgrowth (SIBO) for 21 days. Individuals will return for safety checks every week during the 21-day period. At 21-days, plaque samples and a gingival biopsy will be collected. For diseased individuals SRP will initiate during the 21-day visit at the SIBO quadrant. Visit 6 (28 days) will include the post-biopsy follow up, prophylaxis (for healthy individuals) and SRP (diseased individuals). Subjects receiving SRP may have 2 additional visits (visit 7 at day 35 and visit 8 at day 42) for completing the SRP of all quadrants and will be dependent on individual need. Medical histories, demographics, height and weight, clinical and biological data described above will be recorded and stored on a secure server located at the University of North Carolina. Each participant enrolled into the study will have a unique identification number that has been stripped of any information that could be used by non-study members to identify the subject.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have read, understood and signed an informed consent form.
* Subjects must be able and willing to follow study procedures and instructions.
* Subjects must be adult males or females with a minimum of 18 years (inclusive).
* Subjects must present with at least 20 teeth in the functional dentition, excluding third molars.
* Subjects must have at least 3 teeth in each posterior sextant
* Subjects must be in good general health
* Subjects must be in the healthy (PPC-A) or severe periodontitis (PPC-G) categories according to the PPC (1)

Exclusion Criteria:

* If the sextants identified for the analysis has implants
* All individuals who meet criteria for anti-infective prophylaxis prior to dental procedures
* Chronic disease with oral manifestations including diabetes mellitus.
* Current smoker or one that has stopped smoking less than 2 years prior to enrollment.
* Gross oral pathology other than the periodontal disease.
* Treatment with antibiotics for any medical or dental condition within 1 month prior to the screening examination.
* Chronic treatment (i.e., two weeks or more) with any medication known to affect periodontal status (e.g., phenytoin, calcium antagonists, cyclosporin, coumadin, non-steroidal anti-inflammatory drugs, aspirin) within one month of the screening examination.
* Ongoing medications initiated less than three months prior to enrollment (i.e., medications for chronic medical conditions must be initiated at least three months prior to enrollment).
* Significant organ disease including impaired renal function, heart murmur, history of rheumatic fever or valvular disease, or any bleeding disorder.
* Individuals with prosthetic material used for intra-cardiac repair (e.g. for congenital heart disease), or intra-cardiac devices, cardiac transplant, infective endocarditis and individuals who have had previous infectious complications of prosthetic joint infections
* Infectious diseases such as hepatitis, HIV or tuberculosis.
* Anemia or other blood dyscrasias.
* Anticoagulant therapy or drugs, such as heparin or warfarin.
* Severe unrestored caries, or any condition that is likely to require antibiotic treatment over the trial.
* Pregnant, or expect to become pregnant within the next several months.
* Females of child-bearing capacity must be willing to have pregnancy test to confirm they are not pregnant.
* Females of child-bearing capacity not using any form of contraceptive methods
* Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie T Marchesan, DDS, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB) and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: 9-36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Groups:
- Periodontal Profile Class (PPC-A/PPC-B): Periodontally healthy participants (PPC-A) and mild disease (PPC-B) will wear customized acrylic mouthguard only during tooth brushing for 21 days.
  Customized acrylic mouthguard: Customized acrylic mouthguards extended to cover approximately 2 mm over gingival margins will be fabricated for each subject. Stents will form a seal and rest on the gingiva, but will be relieved on the tooth and tissue side except for the occlusal surfaces to avoid disturbing plaque or gingival tissues. Acrylic stents will cover the area in one sextant where no brushing and flossing teeth is to occur for 21 days.
- Periodontal Profile Class (PPC-G/PPC-E): Participants with severe periodontal disease (PPC-G) and posterior disease (PPC-E) will wear customized acrylic mouthguard only during tooth brushing for 21 days.
  Customized acrylic mouthguard: Customized acrylic mouthguards extended to cover approximately 2 mm over gingival margins will be fabricated for each subject. Stents will form a seal and rest on the gingiva, but will be relieved on the tooth and tissue side except for the occlusal surfaces to avoid disturbing plaque or gingival tissues. Acrylic stents will cover the area in one sextant where no brushing and flossing teeth is to occur for 21 days.
Period: Overall Study
Arm/Group | Periodontal Profile Class (PPC-A/PPC-B) | Periodontal Profile Class (PPC-G/PPC-E)
Started | 36 | 33
Completed | 31 | 23
Not Completed | 5 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Periodontal Profile Class (PPC-A/PPC-B) | Periodontal Profile Class (PPC-G/PPC-E) | Total
Number analyzed (Participants) | 36 | 33 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.0 (12.5) | 42.3 (10.6) | 36.9 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 14 | 37
  Male | 13 | 19 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 23 | 26
  Not Hispanic or Latino | 33 | 10 | 43
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 4 | 4 | 8
  White | 25 | 12 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 14 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36 | 33 | 69

OUTCOME MEASURES:

1. Primary Outcome: Change in Absent in Melanoma 2 (AIM2) mRNA Expression Levels
Description: Gingival tissues derived from study participants were evaluated for AIM2 mRNA expression at baseline (experimental timepoint named Day 0) and at 21 days (experimental timepoint named Day 21). Gene expression was evaluated by quantitative reverse transcription polymerase chain reaction (qRT-PCR) and quantified by the delta-delta-CT method.
Time Frame: Baseline (Day 0), Visit 5 (Day 21)
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Periodontal Profile Class (PPC-A/PPC-B) | Periodontal Profile Class (PPC-G/PPC-E)
Number analyzed (Participants) | 31 | 23
fold change | 0.37 (1.56) | 0.65 (3.29)
Statistical Analysis 1: Comparison: Periodontal Profile Class (PPC-A/PPC-B) vs Periodontal Profile Class (PPC-G/PPC-E); Test type: Superiority; p = 0.3, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Change in Interferon Gamma Inducible Protein 16 (IFI16) mRNA Expression Levels
Description: Gingival tissues derived from study participants were evaluated for IFI16 mRNA expression at baseline (experimental timepoint named Day 0) and at 21 days (experimental timepoint named Day 21). Gene expression was evaluated by qRT-PCR and quantified by the delta-delta-CT method.
Time Frame: Baseline (Day 0), Visit 5 (Day 21)
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Periodontal Profile Class (PPC-A/PPC-B) | Periodontal Profile Class (PPC-G/PPC-E)
Number analyzed (Participants) | 31 | 23
fold change | 0.07 (0.53) | 0.10 (0.61)
Statistical Analysis 1: Comparison: Periodontal Profile Class (PPC-A/PPC-B) vs Periodontal Profile Class (PPC-G/PPC-E); Test type: Superiority; p = 0.5, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Change in the Percentage of AIM2 Positive Cells
Description: Gingival tissues derived from study participants were evaluated for AIM2 immunohistochemical staining at baseline (experimental timepoint named Day 0) and at 21 days (experimental timepoint named Day 21). Cell positivity at baseline and Day 21 was measured by H-score, which consists of (percent low positive cells x 1) + (percent positive cells x 2) + (percent high positive cells x 3).
Time Frame: Baseline (Day 0), Visit 5 (Day 21)
Measure: Mean (Standard Deviation); unit: percent positive cells
Arm/Group | Periodontal Profile Class (PPC-A/PPC-B) | Periodontal Profile Class (PPC-G/PPC-E)
Number analyzed (Participants) | 31 | 23
percent positive cells | -0.71 (29.77) | 4.55 (38.78)
Statistical Analysis 1: Comparison: Periodontal Profile Class (PPC-A/PPC-B) vs Periodontal Profile Class (PPC-G/PPC-E); Test type: Superiority; p = 0.6, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Change in Percentage of Interferon Gamma Inducible Protein 16 (IFI16) Positive Cells
Description: Gingival tissues derived from study participants were evaluated for IFI16 immunohistochemical staining at baseline (experimental timepoint named Day 0) and at 21 days (experimental timepoint named Day 21). Cell positivity at baseline and Day 21 was measured by H-score, which consists of (percent low positive cells x 1) + (percent positive cells x 2) + (percent high positive cells x 3).
Time Frame: Baseline (Day 0), Visit 5 (Day 21)
Measure: Mean (Standard Deviation); unit: percent positive cells
Arm/Group | Periodontal Profile Class (PPC-A/PPC-B) | Periodontal Profile Class (PPC-G/PPC-E)
Number analyzed (Participants) | 31 | 23
percent positive cells | 0.91 (27.81) | 5.46 (58.63)
Statistical Analysis 1: Comparison: Periodontal Profile Class (PPC-A/PPC-B) vs Periodontal Profile Class (PPC-G/PPC-E); Test type: Superiority; p = 0.5, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Correlation of Changes in Periodontal Pathogens With Changes of AIM2
Description: Correlation between temporal changes in periodontal pathogen levels that are statistically significant between Day 0 and Day 21 were correlated with temporal changes in AIM2 expression using Spearman rank correlation coefficients and corresponding 95% confidence intervals.
Time Frame: Baseline (Day 0), Visit 5 (Day 21)
Population: Pathogens that were not present in significance were not evaluated within a group of participants.
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Periodontal Profile Class (PPC-A/PPC-B) | Periodontal Profile Class (PPC-G/PPC-E)
Number analyzed (Participants) | 31 | 23
correlation coefficient
  Prevotellaceae: number analyzed (Participants) | 31 | 0
  Prevotellaceae | -0.1 [-0.47 to 0.29] |
  Bulleidia: number analyzed (Participants) | 31 | 0
  Bulleidia | -0.1 [-0.4 to 0.2] |
  Pseudoramibacter: number analyzed (Participants) | 31 | 0
  Pseudoramibacter | -0.2 [-0.58 to 0.15] |
  Haemophilus: number analyzed (Participants) | 31 | 0
  Haemophilus | 0.28 [-0.1 to 0.6] |
  Gracilibacteria: number analyzed (Participants) | 31 | 0
  Gracilibacteria | 0.3 [-0.05 to 0.6] |
  Alloprevotella: number analyzed (Participants) | 31 | 0
  Alloprevotella | -0.16 [-0.52 to 0.24] |
  Colibacter: number analyzed (Participants) | 31 | 0
  Colibacter | 0.01 [-0.37 to 0.4] |
  Saccharibacteria: number analyzed (Participants) | 31 | 0
  Saccharibacteria | -0.04 [-0.4 to 0.3] |
  Erysipelotrichaceae: number analyzed (Participants) | 31 | 0
  Erysipelotrichaceae | -0.01 [-0.4 to 0.3] |
  Mollicutes: number analyzed (Participants) | 0 | 23
  Mollicutes |  | 0.05 [-0.4 to 0.5]
  Scardovia: number analyzed (Participants) | 0 | 23
  Scardovia |  | -0.01 [-0.4 to 0.4]
  Peptostreptococcaceae: number analyzed (Participants) | 0 | 23
  Peptostreptococcaceae |  | -0.09 [-0.5 to 0.3]
  Stomatobaculum: number analyzed (Participants) | 0 | 23
  Stomatobaculum |  | -0.2 [-0.6 to 0.2]
  Cryptobacterium: number analyzed (Participants) | 0 | 23
  Cryptobacterium |  | -0.17 [-0.5 to 0.2]
  Lautropia: number analyzed (Participants) | 0 | 23
  Lautropia |  | 0.2 [0.2 to 0.6]

6. Secondary Outcome: Correlation of Changes in Periodontal Pathogens With Changes of IFI16
Description: Correlation between temporal changes in periodontal pathogen levels that are statistically significant between Day 0 and Day 21 were correlated with temporal changes in IFI16 expression using Spearman rank correlation coefficients and corresponding 95% confidence intervals.
Time Frame: Baseline (Day 0), Visit 5 (Day 21)
Population: Pathogens that were not present in significance were not evaluated within a group of participants.
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Periodontal Profile Class (PPC-A/PPC-B) | Periodontal Profile Class (PPC-G/PPC-E)
Number analyzed (Participants) | 31 | 23
correlation coefficient
  Prevotellaceae: number analyzed (Participants) | 31 | 0
  Prevotellaceae | -0.3 [-0.6 to 0.06] |
  Bulleidia: number analyzed (Participants) | 31 | 0
  Bulleidia | -0.3 [-0.6 to 0.05] |
  Pseudoramibacter: number analyzed (Participants) | 31 | 0
  Pseudoramibacter | -0.36 [-0.5 to 0.2] |
  Haemophilus: number analyzed (Participants) | 31 | 0
  Haemophilus | 0.4 [-0.008 to 0.6] |
  Gracilibacteria: number analyzed (Participants) | 31 | 0
  Gracilibacteria | 0.2 [-0.2 to 0.5] |
  Alloprevotella: number analyzed (Participants) | 31 | 0
  Alloprevotella | -0.2 [-0.5 to 0.1] |
  Colibacter: number analyzed (Participants) | 31 | 0
  Colibacter | -0.1 [-0.5 to 0.2] |
  Saccharibacteria: number analyzed (Participants) | 31 | 0
  Saccharibacteria | -0.01 [-0.4 to 0.3] |
  Erysipelotrichaceae: number analyzed (Participants) | 31 | 0
  Erysipelotrichaceae | -0.14 [-0.5 to 0.2] |
  Mollicutes: number analyzed (Participants) | 0 | 23
  Mollicutes |  | -0.3 [-0.6 to 0.1]
  Scardovia: number analyzed (Participants) | 0 | 23
  Scardovia |  | -0.18 [-0.5 to 0.2]
  Peptostreptococcaceae: number analyzed (Participants) | 0 | 23
  Peptostreptococcaceae |  | -0.02 [-0.4 to 0.4]
  Stomatobaculum: number analyzed (Participants) | 0 | 23
  Stomatobaculum |  | -0.3 [-0.6 to 0.1]
  Cryptobacterium: number analyzed (Participants) | 0 | 23
  Cryptobacterium |  | -0.25 [-0.6 to 0.2]
  Lautropia: number analyzed (Participants) | 0 | 23
  Lautropia |  | 0.29 [-1.7 to 0.6]

ADVERSE EVENTS:
Time Frame: From the time of informed consent through study completion, up to 56 days.
Arm/Group | Periodontal Profile Class (PPC-A/PPC-B) | Periodontal Profile Class (PPC-G/PPC-E)
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/33
Other Adverse Events (participants affected / at risk) | 0/36 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-06): https://cdn.clinicaltrials.gov/large-docs/97/NCT03513497/Prot_SAP_001.pdf
  • Informed Consent Form (2022-09-27): https://cdn.clinicaltrials.gov/large-docs/97/NCT03513497/ICF_000.pdf